CLINICAL TRIAL: NCT06332807
Title: An Open-Label, Multiple-Center, Phase I/II Dose Escalation Study for the Safety and Efficacy of NGGT002 in Adults With Classic Phenylketonuria
Brief Title: AAV Gene Therapy Clinical Study in Adult Classic PKU (PHEdom)
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: NGGT INC. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NGGT002-P-2301
Record Dates: First submitted 2024-02-07; First posted 2024-03-27 (Actual); Last update posted 2025-12-02 (Actual); Status verified 2025-11

CONDITIONS: Phenylketonurias
Keywords: PAH; Phenylalanine; Phenylalanine Hydroxylase
MeSH Terms: conditions — Phenylketonurias

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- NGGT002 (Experimental): Low dose and high dose group:
  Six to twelve patients will be enrolled into two cohorts at two dose levels. The safety of this study can be ensured by selecting the highest dose under the No Observed Adverse Effect Level (NOAEL) doses observed in preclinical toxicology studies.
  Interventions: Genetic: NGGT002

INTERVENTIONS:
Genetic: NGGT002 — adeno-associated viral vector with human phenylalanine hydroxylase gene

SUMMARY:
This is a Phase 1/2, open-label, multiple-center, dose escalation and cohort expansion study to evaluate the safety and efficacy of NGGT002 in adult subjects with classic Phenylketonuria (PKU). NGGT002 is an rAAV8 based vector carrying a functional copy of the human PAH gene.

Participants will receive a single administration of NGGT002 and will be followed for safety and efficacy for 5 years.

DETAILED DESCRIPTION:
This study will evaluate the safety and efficacy of NGGT002 gene therapy with two dose cohorts in adult subjects with diagnosis of classic PKU, a condition characterized by severe PAH deficiency with no residual enzyme activity. NGGT002 will be administered through intravenous infusion. In Part 1 of the study, subjects will receive NGGT002 at the low dose. Dosing of the first 3 subjects will be staggered. Following evaluation of data from the first 3 subjects, a decision can be made to either escalate to the high dose level or expand the low dose cohort with additional 3 subjects. Upon completion of Part 1 study, based on the evaluation of and safety and efficacy, the study may be stopped or proceed to Part 2. In Part 2, the same process will be conducted with 3 -6 subjects dosed at the high dose.

ELIGIBILITY:
Inclusion Criteria:

1. Is willing and able to provide written, signed informed consent after the nature of the study has been explained and prior to any research-related procedures; a legally authorized representative may provide written consent and assent may be requested.
2. Male and female subjects with diagnosis of classic PKU, a condition characterized by severe PAH deficiency with confirmed PAH mutations predicted with no residual enzyme activity. A list of PAH mutations for classic PKU based on in vitro PAH activity (Himmelreich et al., 2018) and the genotype-phenotype correlation (Garbade et al., 2019) can be found in BIOPKU genotypes database (http://www.biopku.org/pah).
3. Adults aged 18-55 at the time of informed consent
4. Subjects intolerant or unresponsive to available medical therapies, such as Kuvan, Playnzip, etc.
5. Subjects who have been on medications, such as Kuvan, Palynziq, etc but have come off for medical reasons or the patient's decision at least 28 days prior to signing the consent form (Subjects who have good disease control on these existing therapies will not be included in this study).
6. At least 1 documented measurements of Phe ≥ 600 μmol/L while on usual diet in the preceding 6 months.
7. Subjects are willing to record their diet and follow the instruction of dietitians during the trial.
8. Willingness and capable per Investigator opinion to comply with study procedures and requirements.
9. Women of child bearing potential must be confirmed as negative non pregnant subjects by blood pregnancy test from day -28 to day 0. Subjects must agree to use a highly effective form of contraception from the time of NGGT002 administration until a minimum of 1 year after NGGT002 administration, and for male subjects, a minimum of 3 consecutive semen samples are negative for AAV8 after administration of NGGT002. Highly effective birth control methods include:

   * documented vasectomy or permanent sterilization
   * condom
   * combined (estrogen and progestogen-containing) hormonal contraception (oral, intravaginal or transdermal)
   * progestogen-only hormonal contraception associated with inhibition of ovulation (oral, injectable or implantable)
   * intrauterine device
   * intrauterine hormone-releasing system
   * sexual abstinence is acceptable only as true abstinence and when in line with the preferred and usual lifestyle of the subject. Periodic abstinence (e.g., calendar, ovulation, hypothermal, post-ovulation) is not acceptable as a form of abstinence.

Exclusion Criteria:

1. Subjects with PKU that is not due to PAH mutation
2. Presence of anti-AAV8 neutralizing antibodies
3. Prior to dosing, subjects exceed the limit of any of the following liver function and hematology tests in two consecutive blood laboratory tests:

   * Alanine aminotransferase (ALT) >1.5×ULN and/or aspartate aminotransferase (AST) >1.5×ULN
   * Alkaline phosphatase (ALP) >1.5×ULN
   * Total bilirubin (TBil) >1.5×ULN, direct bilirubin >1.5×ULN
   * International normalized ratio (INR) > 1.5
   * Blood creatinine (Scr) >1.5×ULN
   * Hematology values outside of the normal range (Hemoglobin <110 g/L (male), <100 g/L (female), white blood cell <3.0×10^9/L, neutrophil <1.5×10^9/L, platelet <100×10^9/L)
   * Hemoglobin A1c >6% or fasting glucose >6.1 mmol/L
4. At the time of screening, abnormal vital signs (i.e. Temperature<36.3°C or >37.4°C; Blood pressure<100/60 mmHg or >130/80 mmHg; heart rate <60/min or>100/min; respiratory rate <12/min or >18/min; oxygen saturation<95%), physical examination, laboratory tests, or other related results that have clinical significance, and the researchers believe they are unsuitable for enrollment.
5. Contraindications to corticosteroid use or possible deterioration of corticosteroid use assessed and determined by the Investigator.
6. Active infection with hepatitis A virus (HAV ribonucleic acid [RNA] positive), active or occult hepatitis B virus infection (positive HBV-DNA or anti-HBc positive with negative hBsAg, HBV surface antigen), active infection with hepatitis C virus (HCV RNA positive), infection with the human immunodeficiency virus (HIV) as measured by antibodies to HIV-1 and HIV-2, active or latent infection with tuberculosis (TB) measured by Quantiferon Gold, infection with syphilis by rapid plasma regainn (RPR) and/or serum syphilis antibody, treponema pallidum particle agglutination (TPPA).
7. Subjects with history of liver disease such as clinically significant steatosis, fibrosis, non-alcoholic steatohepatitis (NASH) and cirrhosis, biliary disease within 6 months of informed consent; except for Gilbert's syndrome.
8. All types of past and current malignancy
9. Imaging (liver ultrasound) proved the existence of Liver fibrosis, liver cirrhosis and other serious liver diseases
10. Severe diseases in the cardiovascular, respiratory, digestive tract, endocrine, kidney, blood, nervous, mental and other systems before screening.
11. History of allergy to Albumin (Human)
12. The subjects who have Substance Use Disorder (for example alcohol, heroin, amphetamine, etc)
13. The subjects who have received any gene therapy in the past, regardless of when it was administered.
14. The subjects who have received any investigational treatment and took drugs within 3 months before screening (or 5 half-lives, if longer)
15. Subjects with elevated circulating serum alpha-fetoprotein (AFP)
16. Other conditions that the Investigators deemed inappropriate for enrollment, such as PKU severe comorbidities and conditions (i.e. renal insufficiency or kidney failure, osteoporosis, anemia, acid reflux or gastro-esophageal ulcer, major depression, epilepsy, etc.), which may be deteriorated with the potential risks of NGGT002.
17. Subjects who are presently on available medications for the treatment of PKU, such as Kuvan, Palynziq, etc.
18. Subjects who weight over 120 Kg
19. Subjects who consume too much natural protein (>2 g/Kg body weight/day) in their daily diet
20. Breastfeeding subjects will not be included in the study

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 12 (Estimated)
Dates: Start 2025-01-10 (Actual); Primary Completion 2030-12-30 (Estimated); Study Completion 2030-12-30 (Estimated)

PRIMARY OUTCOMES:
Incidence and severity of Adverse Events (AEs) | Baseline to Week 52 and during Year 1 to 5
  Incidence and severity of AEs, including serious AEs (SAEs) as assessed by CTCAE v5.0 of a single administration of NGGT002.
Change from baseline in clinical laboratory values | Baseline to Week 52 and during Year 1 to 5
  Change in chemistry values including liver function tests, hematology and urinalysis.
Change from baseline in 12-lead electrocardiograms (ECGs), vital signsand physical examinations | Baseline to Week 52 and during Year 1 to 5
  Subjects change from baseline in 12-lead electrocardiograms (ECGs), vital signs and physical examinations.
Change from baseline in Plasma Phe Concentration | Baseline to Week 52 and during Year 1 to 5
  To evaluate the efficacy in change of plasma Phe concentration of IV infusion of NGGT002 in adults with classic PKU at Week 12, Week 28, Week 52 and during Year 1 to 5.

SECONDARY OUTCOMES:
Incidence of sustained plasma Phe concentration of ≤360 μmol/L (6 mg/dL) at Week 12, Week 28, Week 52 and during Year 1 to 5 post dose | Baseline to Week 52 and during Year 1 to 5
  Subjects achieving a sustained plasma Phe concentration ≤360 μmol/L (6 mg/dL) at Week 12, Week 28, Week 52 and during Year 1 to 5 post dose.
Change from baseline in total protein intake at at Week 28, Week 52 and during Year 1 to 5 post dose | Baseline to Week 52 and during Year 1 to 5
  Subject achieving a change from baseline in total protein intake at Week 28, Week 52 and during Year 1 to 5 post dose.
Change in Phenylketonuria Quality of Life Questionnaire (PKU-QOL) | Baseline to Week 52 and during Year 1 to 5
  Change in PKU-QOL at Week 28, Week 52 and during Year 1 to 5 post dose.

CONTACTS AND LOCATIONS:
Locations (5):
- United States (5):
  - Children's Hospital of Orange County Hospital, Orange, California
  - University of Minnesota, Minneapolis, Minnesota
  - Atlantic Health System, Morristown, New Jersey
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - University or Texas, Southwestern medical Center, Dallas, Texas

IPD SHARING:
Plan to Share IPD: No